CLINICAL TRIAL: NCT06273163
Title: Identifying Strategies to Curtail Weight Regain After GLP-1 Receptor Agonist Treatment Cessation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended, unable to reach recruitment goal.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: UT Southwestern Nutrition Obesity Research Center (Unknown)
Responsible Party: Principal Investigator, Kelseanna Hollis-Hansen, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STU-2023-1168
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Obesity
Keywords: Glucagon-Like Peptide-1 Receptor Agonists; Body Weight Maintenance
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Randomized repeated measures between-subjects design
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Complete masking is not feasible given the nature of the interventions - the program coordinator and participants will know if the participant receives home delivered medically tailored meals, a smart device application subscription, or usual care. The care provider will not be told the participants group assignment, but the participant may reveal it themselves in discussions with the provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medically tailored meals (Experimental): Participants will receive 10 medically tailored meals per week (40 meals per month) for four-months.
  Interventions: Other: Medically tailored meals; Other: Usual care
- Noom® (Experimental): Participants will receive a paid Noom® subscription for four-months. Noom® is a subscription-based mobile application that provides food intake and exercise tracking and uses principles from psychology to motivate behavior change.
  Interventions: Behavioral: Noom®; Other: Usual care
- Usual care (Placebo Comparator): Participants will receive usual care from their provider.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Medically tailored meals — Medically tailored meals are nutritious meals formulated for weight wellness.
  Arms: Medically tailored meals
Behavioral: Noom® — Noom® is a subscription-based mobile application used to support healthy eating and exercise behavior change.
  Arms: Noom®
Other: Usual care — Care is provided at the discretion of the individual provider (e.g., usual care).

SUMMARY:
Longitudinal studies show there is a steep increase in weight regain in the first 3-4 months after stopping GLP-1 receptor agonist medications (GLP-1s) and most patients regain most of their weight within a year. Insurers now question the utility of GLP-1s for weight loss as they are hesitant to cover these costs long-term (~$833 per person per month). Some patients would also prefer not to take these medications in perpetuity and are likely to struggle with lifelong adherence. These challenges present an opportunity to test alternative interventions, such as meal replacements and behavioral treatments, to support weight maintenance after successful weight loss with GLP-1s. This regimen would allow patients to benefit from significant weight loss in the first year of taking GLP-1s and use more cost effective and sustainable strategies for long-term maintenance.

DETAILED DESCRIPTION:
In the proposed study the investigators will execute a pilot randomized controlled trial to identify whether medically tailored meals (MTM, Group 1, N=20) and/or Noom®, a mobile application (Group 2, N=20) are associated with greater treatment adherence and satisfaction than usual care (Group 3, N=20) after GLP-1 Receptor Agonist cessation. The investigators will enroll adults 18 and older that have lost more than 10% of their bodyweight taking GLP-1 Receptor Agonist and ceased treatment within the past 30-days. For four-months, Group 1 will receive 40 MTM per month, Group 2 will receive a Noom® subscription, and Group 3 will receive lifestyle counseling per standard of care.

ELIGIBILITY:
Inclusion criteria:

* 18 years of age or older;
* ability to read, write, and speak English;
* ability to provide informed consent;
* greater than 10% GLP-1 Receptor Agonist induced weight loss
* less than 30-days since GLP-1 Receptor Agonist cessation;
* willing to participate.

Exclusion criteria:

* major psychiatric illness or substance misuse that could impair ability to participate;
* presence of a medical condition or dietary restriction precluding eating study meals or weight loss (e.g., medical condition requiring liquid diet, pregnancy, eating disorder);
* participation in a study or program involving medically tailored meals or Noom® within the past 12-months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Intervention Adherence | 4-months
  Adherence will be measured using the Perceived Behavior subscale (6-items) from the validated Treatment Adherence Perception Questionnaire (TAPQ).
Intervention Satisfaction | 4-months
  The Abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9) will be used to measure satisfaction, and be adapted for the interventions understudy. Responses are provided on a 7-point Likert scale ranging from extremely satisfied to extremely dissatisfied. Scores are then transformed to a 0-100 scale with a higher score indicating greater treatment satisfaction.

SECONDARY OUTCOMES:
Percent weight loss maintained | 4-months
  The electronic health record will be used to determine the participants' weight prior to and at the end of GLP-1 Receptor Agonist treatment to determine the percent of bodyweight lost on GLP-1 Receptor Agonist. Weight will be measured using a Bluetooth scale pre- and post-intervention to calculate the percent of weight loss maintained at the end of the study.
Diet quality | 4-months
  Healthy eating index-2015 (HEI-2015), scored according to National Cancer Institute (NCI) guidelines from 0-100, with 0 indicating no intake of nutritious foods and 100 indicating higher intake of nutritious food.

OTHER OUTCOMES:
Incremental cost effective ratio (ICER) | 4-months
  Incremental cost effectiveness ratios (ICER) will be calculated as the difference in cost to implement each intervention divided by 1) the increase in HEI score and 2) percent weight loss maintained.

CONTACTS AND LOCATIONS:
Overall Officials: Kelseanna Hollis-Hansen, PhD, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided